CLINICAL TRIAL: NCT00460798
Title: A Non-Interventional Study With SUTENT® In The First Line Treatment Of Renal Cell Cancer
Brief Title: SUTENT® In The First Line Treatment Of Renal Cell Carcinoma
Acronym: SUNIKA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Other Study IDs: A6181115
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Sunitinib; kidney diseases; urogenital neoplasms; kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Diseases; Urogenital Neoplasms; Kidney Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-Interventional Study
  Interventions: Other: Sutent: observational study

INTERVENTIONS:
Other: Sutent: observational study — SUNIKA - A Non-Interventional Study With SUTENT® In The First Line Treatment Of Renal Cell Carcinoma
  Other Names: sunitinib malate

SUMMARY:
This non-interventional study includes patients with advanced and/or metastatic renal cell carcinoma who are treated with SUTENT and who did not receive any other systemic therapy before. The aim of the trial is to increase knowledge about quality of life, safety, efficacy and tolerability under conditions of routine use of Sutent. The individual observation period of each patient will be

1 year.

DETAILED DESCRIPTION:
The Statistical Analysis Plan provides detailed specification of the analysis

ELIGIBILITY:
Inclusion Criteria:

* First-line treatment in patients with metastatic renal cell carcinoma

Exclusion Criteria:

* Any previous systemic therapy of renal cell carcinoma except for adjuvant treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated by office-based oncologists, office-based urologists specialized in oncology or hospital-based oncologist/urologists
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181115&StudyName=SUTENT%AE%20In%20The%20First%20Line%20Treatment%20Of%20Renal%20Cell%20Carcinoma%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 448 subjects were enrolled. Subjects were eligible for treatment analysis if complete dosing data were available. Of the total 448 subjects enrolled, 421 were eligible for treatment analysis and were recorded as treated. Three subjects who were included in analysis had missing demographic data.
Groups:
- Sunitinib: Sunitinib malate (Sutent) was administered and dosed as stipulated in the Summary of Product Characteristics (SmPC) and was used solely in accordance with the medical and therapeutic needs. The recommended dose of Sutent was 50 mg once daily, administered orally over 4 weeks, followed by a rest period of 2 weeks (4/2 regimen). One treatment cycle = 6 weeks.
Period: Overall Study
Arm/Group | Sunitinib
Started | 448
Treated | 421 (Subjects with complete dosing information were recorded as 'Treated')
Completed | 108
Not Completed | 340
Not completed — Death | 59
Not completed — Adverse Event | 27
Not completed — Lost to Follow-up | 19
Not completed — Progressive Disease | 99
Not completed — Other | 27
Not completed — Ongoing at Date of Cut-Off | 82
Not completed — Missing/Incomplete Dosing Information | 27

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 418
Age, Customized [Number; unit: Participants]
  18 to 44 Years | 12
  45 to 64 Years | 148
  >=65 Years | 256
  Unspecified | 2
Sex/Gender, Customized [Number; unit: Participants]
  Male | 314
  Female | 103
  Unspecified | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Categorical Best Overall Response
Description: Best overall reponse based on investigator's disease status assessment. Complete response(CR)=disappearance of all target lesions.Partial Response(PR)=≥30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions.Progressive disease(PD)=≥20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of longest dimensions since treatment start or appearance of ≥1 new lesions. Stable disease(SD)=neither shrinkage for PR or increase for PD taking as reference smallest sum of longest dimensions since treatment start.
Time Frame: Start of Treatment up through 12 Months or Early Discontinuation
Population: Full Analysis Set (FAS) = All participants who had taken at least 1 dose of study medication and had a post baseline efficacy measurement
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 352
Participants
  Complete Response (CR) | 13
  Partial Response (PR) | 130
  Stable Disease/No Response | 120
  Progressive Disease (PD) | 58
  Indeterminate | 31
Statistical Analysis 1: Comparison: Sunitinib; Objective Response Rate (ORR) = Percentage of participants with best overall response of CR or PR; Test type: Superiority or Other; Obective Response Rate (Percent) = 40.6, 95% CI 2-sided [35.5 to 46.0] — Exact method based on binomial distribution

2. Primary Outcome: Number of Participants With Objective Response
Description: Objective response (CR or PR) based on investigator's overall objective tumor assessment at final visit according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as disappearance of all target lesions. PR was defined as a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: 12 Months or Early Discontinuation
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 352
Participants | 77

3. Primary Outcome: Time to Progression (TTP)
Description: TTP = time from date of first dose to date of first recording of PD. Participants who did not have a recorded PD at any of the visits or at Overall Objective Tumor Assessment at 12 months were treated as censored at the date of the last available follow up for disease response/tumor assessment.
Time Frame: Start of Treatment up through 12 Months or Early Discontinuation
Population: FAS. Number of participants with progression = 162; Number of participants censored = 190
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 352
Months | 12.0 [10.3 to 13.5]

4. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG performance status measured on 6 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all self care, unable to carry out any work activities; 3=Capable of only limited self care, confined to bed/chair >50% of waking hours; 4=Completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=Dead. 0=Best status, 5=Worst status
Time Frame: Baseline, 3, 6, 9 and 12 Months
Population: FAS. ECOG performance status data was not reported for 24, 32, 96, 174, and 174 participants at baseline, 3, 6, 9, and 12 months, respectively.
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 352
Participants
  Fully Active (Baseline) | 84
  Restricted Physical Strenuous Activity (Baseline) | 179
  Capable of Self Care Only (Baseline) | 58
  Capable of Limited Self Care Only (Baseline) | 6
  Completely Disabled (Baseline) | 1
  Fully Active (3 Months) | 57
  Restricted Physical Strenuous Activity (3 Months) | 169
  Capable of Self Care Only (3 Months) | 78
  Capable of Limited Self Care Only (3 Months) | 13
  Completely Disabled (3 Months) | 3
  Fully Active (6 Months) | 43
  Restricted Physical Strenuous Activity (6 Months) | 137
  Capable of Self Care Only (6 Months) | 55
  Capable of Limited Self Care Only (6 Months) | 18
  Completely Disabled (6 Months) | 2
  Dead (6 Months) | 1
  Fully Active (9 Months) | 31
  Restricted Physical Strenuous Activity (9 Months) | 103
  Capable of Self Care Only (9 Months) | 30
  Capable of Limited Self Care Only (9 Months) | 9
  Completely Disabled (9 Months) | 4
  Dead (9 Months) | 1
  Fully Active (12 Months) | 27
  Restricted Physical Strenuous Activity (12 Months) | 88
  Capable of Self Care Only (12 Months) | 46
  Capable of Limited Self Care Only (12 Months) | 7
  Completely Disabled (12 Months) | 6
  Dead (12 Months) | 4

5. Primary Outcome: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Scores
Description: EORTC QLQ-C30: 5 functional scales (physical, role, cognitive, emotional, and social), a global health status/quality of life (QoL) scale, 3 symptom scales (nausea and vomiting, pain, fatigue) and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties). All scales and single-item measures range=0 to 100. High score for a functional scale=high/healthy level of functioning. High score for global health status/QoL=high QoL. High score for symptom scale/single item=high level of symptomatology/problems
Time Frame: Baseline, 3, 6, 9 and 12 Months
Population: FAS. n=number of participants with EORTC scale score data available at each specified time point
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 352
Scores on Scale
  Global Health Status/QoL (Baseline), (n=213) | 53.9 (22.16)
  Global Health Status/QoL (3 Months), (n=195) | 54.7 (20.52)
  Global Health Status/QoL (6 Months), (n=144) | 54.3 (21.07)
  Global Health Status/QoL (9 Months), (n=82) | 56.4 (20.34)
  Global Health Status/QoL (12 Month), (n=80) | 54.5 (20.75)
  Physical Functioning (Baseline), (n=212) | 70.0 (24.21)
  Physical Functioning (3 Months), (n=192) | 67.4 (24.53)
  Physical Functioning (6 Months), (n=144) | 68.3 (23.68)
  Physical Functioning (9 Months), (n=81) | 68.8 (19.37)
  Physical Functioning (12Months), (n=79) | 67.3 (23.54)
  Role Functioning (Baseline), (n=208) | 58.3 (31.98)
  Role Functioning (3 Months), (n=193) | 54.2 (31.79)
  Role Functioning (6 Months), (n=143) | 56.5 (30.26)
  Role Functioning (9 Months), (n=84) | 56.7 (26.65)
  Role Functioning (12Months), (n=80) | 55.0 (27.23)
  Emotional Functioning (Baseline), (n=215) | 61.5 (26.55)
  Emotional Functioning (3 Months), (n=194) | 60.9 (26.78)
  Emotional Functioning (6 Months), (n=144) | 65.1 (24.01)
  Emotional Functioning (9 Months), (n=84) | 66.7 (21.49)
  Emotional Functioning (12 Months), (n=80) | 65.5 (24.22)
  Cognitive Functioning (Baseline), (n=215) | 78.8 (24.81)
  Cognitive Functioning (3 Months), (n=193) | 74.0 (26.94)
  Cognitive Functioning (6 Months), (n=144) | 75.1 (22.30)
  Cognitive Functioning (9 Months), (n=84) | 75.8 (19.43)
  Cognitive Functioning (12 Months), (n=80) | 72.7 (25.19)
  Social Functioning (Baseline), (n=214) | 65.3 (31.02)
  Social Functioning (3 Months), (n=194) | 61.7 (31.80)
  Social Functioning (6 Months), (n=143) | 64.8 (30.07)
  Social Functioning (9 Months), (n=82) | 72.2 (25.40)
  Social Functioning (12 Months), (n=79) | 64.1 (29.97)
  Fatigue (Baseline), (n=214) | 42.5 (27.73)
  Fatigue (3 Months), (n=194) | 49.1 (27.60)
  Fatigue (6 Months), (n=144) | 45.4 (26.17)
  Fatigue (9 Months), (n=84) | 43.4 (25.91)
  Fatigue (12 Months), (n=80) | 44.3 (26.01)
  Nausea and Vomiting (Baseline), (n=214) | 12.3 (20.85)
  Nausea and Vomiting (3 Months), (n=194) | 16.2 (20.39)
  Nausea and Vomiting (6 Months), (n=144) | 14.4 (18.24)
  Nausea and Vomiting (9 Months), (n=84) | 14.3 (21.04)
  Nausea and Vomiting (12 Months), (n=80) | 14.0 (19.57)
  Pain (Baseline), (n=214) | 33.6 (33.00)
  Pain (3 Months), (n=193) | 32.0 (30.47)
  Pain (6 Months), (n=144) | 32.5 (31.12)
  Pain (9 Months), (n=84) | 31.7 (29.91)
  Pain (12 Months), (n=80) | 34.4 (25.89)
  Dyspnoea (Baseline), (n=214) | 30.8 (31.71)
  Dyspnoea (3 Months), (n=194) | 32.0 (30.13)
  Dyspnoea (6 Months), (n=144) | 26.2 (27.07)
  Dyspnoea (9 Months), (n=84) | 25.0 (24.75)
  Dyspnoea (12 Months), (n=80) | 29.6 (29.53)
  Insomnia (Baseline), (n=213) | 30.8 (33.24)
  Insomnia (3 Months), (n=192) | 33.0 (32.71)
  Insomnia (6 Months), (n=144) | 31.3 (31.09)
  Insomnia (9 Months), (n=84) | 28.2 (30.83)
  Insomnia (12 Months), (n=80) | 31.3 (33.27)
  Appetite Loss (Baseline), (n=214) | 27.7 (34.18)
  Appetite Loss (3 Months), (n=194) | 36.3 (35.55)
  Appetite Loss (6 Months), (n=144) | 34.5 (33.31)
  Appetite Loss (9 Months), (n=84) | 32.1 (34.50)
  Appetite Loss (12 Months), (n=80) | 28.8 (32.15)
  Constipation (Baseline), (n=214) | 12.6 (24.21)
  Constipation (3 Months), (n=194) | 13.4 (24.54)
  Constipation (6 Months), (n=144) | 12.7 (24.62)
  Constipation (9 Months), (n=83) | 11.2 (23.44)
  Constipation (12 Months), (n=80) | 8.3 (18.75)
  Diarrhoea (Baseline), (n=214) | 10.4 (23.07)
  Diarrhoea (3 Months), (n=194) | 27.1 (30.47)
  Diarrhoea (6 Months), (n=144) | 28.0 (29.41)
  Diarrhoea (9 Months), (n=84) | 32.1 (32.91)
  Diarrhoea (12 Months), (n=80) | 37.5 (35.33)
  Financial Difficulties (Baseline), (n=212) | 19.2 (30.08)
  Financial Difficulties (3 Months), (n=193) | 19.7 (29.92)
  Financial Difficulties (6 Months), (n=143) | 21.9 (29.10)
  Financial Difficulties (9 Months), (n=82) | 20.7 (29.92)
  Financial Difficulties (12 Months), (n=79) | 24.1 (30.16)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 100/421
Other Adverse Events (participants affected / at risk) | 232/421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=421)
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal symptom (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Oesophagitis (Gastrointestinal disorders) | 2
Small intestinal perforation (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Death (General disorders) | 2
Disease progression (General disorders) | 8
Gait disturbance (General disorders) | 2
General physical health deterioration (General disorders) | 3
Multi-organ failure (General disorders) | 1
Pain (General disorders) | 2
Sudden cardiac death (General disorders) | 3
Ulcer haemorrhage (General disorders) | 1
Acute hepatic failure (Hepatobiliary disorders) | 1
Gallbladder perforation (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Bronchopneumonia (Infections and infestations) | 2
Conjunctivitis infective (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Postoperative wound infection (Infections and infestations) | 1
Ear injury (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 2
Haemoglobin abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 3
Renal failure chronic (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 2
Infarction (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=421)
Anaemia (Blood and lymphatic system disorders) | 20
Anaemia of malignant disease (Blood and lymphatic system disorders) | 2
Bicytopenia (Blood and lymphatic system disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 17
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 22
Angina pectoris (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Epidermolysis (Congenital, familial and genetic disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 7
Eyelid oedema (Eye disorders) | 3
Lacrimation increased (Eye disorders) | 2
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 10
Abdominal wall disorder (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Anal pruritus (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 64
Diverticulum (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 15
Eructation (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Gastric disorder (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 2
Glossodynia (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 43
Oesophageal pain (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Painful defaecation (Gastrointestinal disorders) | 1
Rectal prolapse (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 2
Retching (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 30
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 20
Adverse event (General disorders) | 1
Asthenia (General disorders) | 4
Chest pain (General disorders) | 1
Chills (General disorders) | 3
Death (General disorders) | 1
Disease progression (General disorders) | 1
Face oedema (General disorders) | 2
Fatigue (General disorders) | 37
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 10
Ill-defined disorder (General disorders) | 1
Impaired healing (General disorders) | 1
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 4
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 28
Mucous membrane disorder (General disorders) | 2
Oedema (General disorders) | 6
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 13
Pyrexia (General disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Abscess (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Genital candidiasis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Paronychia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood pressure increased (Investigations) | 4
Blood thyroid stimulating hormone increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 1
Granulocyte count (Investigations) | 1
Haemoglobin (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Muscle enzyme increased (Investigations) | 1
Weight decreased (Investigations) | 4
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Appetite disorder (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Obesity (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ageusia (Nervous system disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 19
Dyskinesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Hemiplegia (Nervous system disorders) | 1
Hypertonia (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 4
Paraplegia (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 5
Food aversion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Genital pain (Reproductive system and breast disorders) | 1
Genital rash (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Blister (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 5
Hair colour changes (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 28
Petechiae (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 5
Skin irritation (Skin and subcutaneous tissue disorders) | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 4
Tooth extraction (Surgical and medical procedures) | 1
Arterial disorder (Vascular disorders) | 1
Blood pressure inadequately controlled (Vascular disorders) | 1
Hyperaemia (Vascular disorders) | 1
Hypertension (Vascular disorders) | 22
Hypotension (Vascular disorders) | 3
Peripheral coldness (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 2
Venous thrombosis limb (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Owing to extent of missing data, the planned TTP analyses derived from standardized lesion measurement was not reported. An additional TTP analysis using Investigator Disease Status and Overall Objective Tumor Assessments at 12 months was reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.